CLINICAL TRIAL: NCT01795872
Title: BENEFIT 11 a Long-term Follow-up Study of the BENEFIT (Betaferon/Betaseron in Newly Emerging Multiple Sclerosis for Initial Treatment, 304747), BENEFIT Follow-up (305207) Studies and BENEFIT Extension (311129) Study to Further Evaluate the Progress of Patients With First Demyelinating Event Suggestive of Multiple Sclerosis
Brief Title: Follow-up Study After 11 Years of Patients Who Were Included in the BENEFIT Trial (304747) With a First Demyelinating Event Suggestive of Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16401; 2012-005262-35 (EudraCT Number)
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Several diagnostic procedures (Other)
  Interventions: Procedure: Several diagnostic procedures

INTERVENTIONS:
Procedure: Several diagnostic procedures — No drug will be assigned, diagnostic assessment within the study.

SUMMARY:
This study assesses clinical and imaging long-term data, after early or delayed interferon-beta-1b treatment in patients with a first demyelinating event suggestive of multiple sclerosis (MS), 11 years after enrollment in the Betaferon/Betaseron in Newly Emerging Multiple Sclerosis for Initial Treatment (BENEFIT) study (304747). The main objectives are to describe the disease course, change in disability, cognitive function, resource use and employment status, in relation to Interferon beta-1b in the long term.

DETAILED DESCRIPTION:
As optic coherence tomography (OCT) and magnetic resonance imaging (MRI) studies are essential to standardize the procedures and assessments for all OCT and MRI test centers that may take part in this study, 122 additional volunteers will be enrolled to test the dummy scans of OCT and MRI, only.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with clinical-isolated syndrome or multiple sclerosis who have been treated at least once in BENEFIT Study 304747

Exclusion Criteria:

* Patients who, according to the investigator's judgment, have medical, psychiatric, or other conditions that compromise the patient's ability to understand the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time to First Relapse by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  Relapses are key features of the clinical presentation of multiple sclerosis. Relapses were assessed retrospectively based on clinical records and subject history. Time to first relapse is the difference from date of first relapse to the date of the BENEFIT baseline visit +1 or time to first relapse is the difference from date of last clinical visit to the date of the BENEFIT baseline visit + 1 (right censored).
Time to Clinically Definite Multiple Sclerosis (CDMS) Represented by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  CDMS could be reached due to a qualifying relapse or sustained progression of 1.5 points on the expanded disability status scale (EDSS) as compared to the lowest EDSS obtained during screening or Day 1 and a total EDSS of >=2.5. The validity of CDMS diagnoses was confirmed by a central committee. The EDSS scale quantifies disability in multiple sclerosis (MS) in 8 functional systems, values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on an ordinal scale. Time to CDMS = the difference from date of CDMS to the date of Day 1 + 1 or time to CDMS = the difference from date of last clinical visit to the Day 1+1 (right censored).
Number of Subjects With Diagnosis of Multiple Sclerosis Within Eleven years after Clinically-Isolated Syndrome (CIS) According to McDonald 2001 and 2010 Criteria | Year 11
  MS according to the criteria by McDonald was reached if, in addition to the single clinical demyelinating event, both dissemination in space (DIS) and dissemination in time (DIT) were established by magnetic resonance imaging (MRI) criteria or a new relapse. Number of subjects with diagnosis of MS within 11 years after CIS according to McDonald 2001 and 2010 criteria were reported.
Disease Course as Assessed at the Time of BENEFIT 11 | Year 11
  Current diagnosis of MS type were categorized with regard to McDonald 2001 and McDonald 2010 criteria were recorded. CIS and silent disease (no relapse, no sustained EDSS progression and no new MRI lesion), McDonald MS not fulfilling the criteria for CDMS, RRMS (CDMS with relapses without evidence for a secondary disease course), SPMS (CDMS with relapses and evidence for a progressive disease course), Revised diagnosis (other reason than MS found for CIS) and Not assessable. Not assessable means McDonald 2001 and McDonald 2010 criteria could not be judged due to missing MRI scan at BENEFIT 11. Number of subjects with current diagnosis of MS at the time of BENEFIT 11 was assessed.
Percentage of Subjects Converting to Secondary Progressive Multiple Sclerosis (SPMS) | Year 11
  SPMS was defined for this study as progressive deterioration observed and sustained for at least 6 months with or without superimposed attacks. Percentage of subjects converting to SPMS were stratified by actual treatment group and baseline EDSS. Baseline EDSS defined as lowest of the EDSS scores obtained during BENEFIT screening or baseline (less than or equal to [<=] median or greater than [>] median).
Time to Secondary Progressive Multiple Sclerosis (SPMS) Represented by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  SPMS was defined for this study as progressive deterioration observed and sustained for at least 6 months with or without superimposed attacks. Time to SPMS was represented by Kaplan-Meier estimates.
Expanded Disability Status Scale (EDSS) at Year 11 | Year 11
  The EDSS scale is a method of quantifying disability in multiple sclerosis in eight functional systems and values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on a scale. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS.
Number of Subjects With Confirmed and Sustained 1-point Expanded Disability Status Scale (EDSS) Progression at Year 11 | Year 11
  The EDSS scale is a method of quantifying disability in multiple sclerosis in eight functional systems and values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on a scale. EDSS progression was defined as an increase in the EDSS of at least 1.0 point compared to initial EDSS score or an increase in the EDSS of at least 1.5 points compared to initial EDSS score, if this score was = 0 points. Confirmed EDSS progression status in any of the previous BENEFIT studies (304747, 305207, 311129) was defined as an EDSS progression observed at two consecutive scheduled visits at least 140 days apart from each other. A confirmed EDSS progression is defined as a confirmed EDSS progression in any of the previous BENEFIT studies or EDSS progression in BENEFIT 11. A sustained EDSS progression is defined as a confirmed EDSS progression in any of the previous BENEFIT studies sustained up to and including the BENEFIT 11 visit.
Number of Subjects With Confirmed 2.5-point Expanded Disability Status Scale (EDSS) Progression at Year 11 | Year 11
  The EDSS scale is a method of quantifying disability in multiple sclerosis in eight functional systems and values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on a scale. EDSS progression was defined as an increase in the EDSS of at least 2.5 points compared to initial EDSS score, if this score was <= 3.5 points, or an increase in the EDSS of at least 2.0 points compared to initial EDSS score, if this score was > 3.5 points. Confirmed EDSS increase status in any of the previous BENEFIT studies (304747, 305207, 311129) was defined as an EDSS increase confirmed at scheduled visits after at least 140 days. A confirmed EDSS increase is defined as a confirmed EDSS increase in any of the previous BENEFIT studies or EDSS increase in BENEFIT 11.
Percentage of Subjects who Ever Reached a Disability Status Scale (DSS) 3 and 6 | Year 11
  The DSS 3, and DSS 6 are important milestones in the course of disability progression and were documented if reached by the subject.
Disability Based Efficacy Domain: Time to Disability Status Scale (DSS) 3 by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  The DSS 3 is an important milestones in the course of disability progression and were documented if reached by the subject. The time point of reaching DSS 3 was obtained retrospectively in the BENEFIT 11 study. Time to respective DSS is the difference between the date of respective DSS and the date of the BENEFIT baseline visit +1. Subjects without event at BENEFIT 11 were censored at the BENEFIT 11 visit. This constituted a right-censored observation. Cumulative probability of reaching DSS 3 at Year 11 were estimated by Kaplan-Meier.
Disability Based Efficacy Domain: Time to Disability Status Scale (DSS) 6 by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  The DSS 6 is an important milestones in the course of disability progression and were documented if reached by the subject. The time point of reaching DSS 6 was obtained retrospectively in the BENEFIT 11 study. Time to respective DSS is the difference between the date of respective DSS and the date of the BENEFIT baseline visit +1. Subjects without event at BENEFIT 11 were censored at the BENEFIT 11 visit. This constituted a right-censored observation. Cumulative probability of reaching DSS 6 at Year 11 were estimated by Kaplan-Meier.
Multiple Sclerosis Functional Composite (MSFC) at Year 11 | Year 11
  The MSFC score consists of three subtests (Timed 25 Foot Walk, 9 Hole Peg Test, 3" Paced Auditory Serial Addition Test [PASAT]) whose Z-standardized results (based on baseline values on Day 1 in Study 304747) were combined into a composite score including upper and lower extremities function, and cognitive function. Standardized results (Z-scores) of the subtests and the overall MSFC Z-score as an average of the three Z-scores were derived using baseline data pooled over both treatment arms as reference population. Higher Z-scores reflect a better neurological status.
Multiple Sclerosis Severity Score (MSSS) at Year 11 | Year 11
  The MSSS added the element of disease duration to the EDSS and was designed to provide a measure of disease severity. It was derived from the EDSS during the data evaluation. The MSSS corrects the EDSS for the duration of disease by using an arithmetical method to compare an individual's disability with the distribution of scores in case of having equivalent disease duration.
Cognitive Function: Paced Auditory Serial Addition Test-3 (PASAT-3) at Year 11 | Year 11
  The Paced Auditory Serial Addition Test (PASAT) is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability.
Cognitive function: Symbol Digit Modalities Test (SDMT) | Year 11
  The Symbol Digit Modalities Test (SDMT) is a cognitive test for sustained attention, concentration, and information-processing speed, with a high sensitivity. Nine different geometrical symbols have one corresponding number each. One-hundred-ten symbols are presented without these numbers; the subject must find the matching number from the top line and verbalize the number to the examiner. The subject is allowed to proceed for 90 seconds, and the number of correct responses in 90 seconds is counted as the total correct score. Also, the numbers of correct responses at 30 and 60 seconds were recorded in this study. Total score ranged from 0 (worst outcome) to best (outcome).
Relapse-Based Efficacy domain: Hazard Ratio for Recurrent Relapses | Year 11
  A relapse was defined as the appearance of a new neurological abnormality or the reappearance of a neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The time to the onset of recurrent relapses was determined for each subject according to the counting process representation for recurrent events. Time to a relapse was right censored if a relapse risk period ended without relapse. Based on the Andersen Gill model the hazard ratio for recurrent relapses was estimated with actual treatment in BENEFIT (304747; i.e. IFNB-1b 250 microgram vs. placebo), steroid use during first event (yes vs. no), onset of disease (multifocal vs. monofocal) and number of T2 lesions on BENEFIT screening MRI (categorized as 2-4, 5-8, >=9) included in the model.
Relapse Based Efficacy Domain: Annualized Relapse Rate | Year 11
  The annualized relapse rate is defined as total number of relapses up to Year 11 divided by the total observation time (last clinical visit minus first day of study treatment administration plus 1 of all subjects) in years.
Time to use of Ambulatory Device Represented by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  Date of use of ambulatory device is defined as the retrospectively obtained time point of first use/dependence. Time to use of ambulatory device is the difference between the date of first use/dependence and the date of the BENEFIT baseline visit +1.
Time to Dependence of Ambulatory Device for Walking Represented by Kaplan-Meier Estimates | Up to Year 11 (Day 3960)
  Date of dependence from ambulatory device is defined as the retrospectively obtained time point of first use/dependence. Time to dependence from ambulatory device is the difference between the date of first use/dependence and the date of the BENEFIT baseline visit +1. Cumulative probability of dependence of ambulatory device for walking represented by Kaplan-Meier estimates at Year 11.
Number of Subjects With Wheelchair Use After 11 years | Year 11

SECONDARY OUTCOMES:
Education Status at Year 11 | Year 11
  Subjects with educational status was categorized as primary school, high school diploma, vocational diploma, collegial studies, university diploma, and missing educational status.
Living Conditions at Year 11 | Year 11
  Subjects living condition were categorized as 'living alone', 'long term care facility', living with spouse, partner, family', 'other' and 'missing'.
Employment Status at Year 11 | Year 11
  Subject's employment status was categorized as 'retired', 'homemaker', 'long term disability', 'employment less than 20 hours (hrs) per week (hrs/week)', employment more than 20 hours per week, 'early retired', 'other', and 'missing'.
Multiple Sclerosis Impact on Employment at Year 11 | Year 11
  Subject's MS impact on employment was categorized as, 'unrelated to MS condition', 'ceased work due to MS', 'never worked', 'reduced working hours', or missing.
Resource Use: Hospitalization During Last 12 months | Year 11
  Hospitalizations were assessed at year 11 only referring to past 12 months. Number of hospitalizations per subject were categorized as, 'none', '1', '2', '3', and '6'.
Resource Use: Visits to Other Specialists During Last 12 months | Year 11
  Visits to Other Specialists were assessed at year 11 only referring to past 12 months. The visits to other specialists were categorized as, 'missing', 'no', 'yes', 'never', and 'unsure'. The other specialists includes, neurologist, nurse clinician, home health aide, visiting nurse, physiotherapist, psychiatrist, psychologist, physician, urologist, social worker and gynecologist.
Resource Use Assessment Questionnaire: Help from Family/Regular Ambulatory Services | Year 11
  Resources use data was assessed cross-sectionally at 11 years. Supportive care was assessed as "assistance given" for the help from family members or friends with "care given" for the number f hors per week needed, as well as "ambulatory services-yes/no" with sub-categories home care, home help, day care center, meals on wheels and child care for the help from professional caregiver.
Resource Use Assessment Questionnaire: Additional Ambulatory Services During Relapse | Year 11
  Resources use data was assessed cross-sectionally at 11 years. Additional ambulatory services during relapse were categorized as, 'missing', 'no', and 'yes'. The additional ambulatory services during relapses were home care, home help, day care center, meals on wheels, and child care.
Resource Use Assessment Questionnaire: Adaptions past 6 months | Year 11
  Resources use data was assessed cross-sectionally at 11 years. The kind of adaptation was categorized as "other part of living", "star lift". "ramps", "alarm", "work", "car", "walking aids", "wheel chair", "spectacles", "special kitchen utensils", "special hygiene utensils", "special writing devices" and " other" with subcategories as 'missing', 'no', and 'yes'.
Patient-Reported Outcomes (PRO)-based Efficacy Domain: Center of Epidemiological Studies Depression Scale (CES-D) Total Score at Year 11 | Year 11
  The CES-D is a measure of depressive symptomatology. The CES-D was a self-administered questionnaire for adults comprising 20 items which evaluated the frequency and severity of depressive symptoms. Subjects were asked to recall the previous 7 days. The total score (0-60) was the sum of the scores of the 20 items. A score of >= 16 suggested a mild to moderate level of depressive symptoms; a score >21 suggested major depressive symptoms.
PRO-based Efficacy Domain: Fatigue Scale for Sensory and Motor Functions (FSMC) | Year 11
  The cognitive and physical fatigue was assessed by the FSMC. The scale comprised of 20 questions (10 items for physical and 10 items for cognitive fatigue) and could be completed within 5 minutes. The items are rated on a 5-point Likert scale (1=does not apply at all to 5=applies completely). The FSMC total score ranges from 20 to 100 where a higher score is associated with a higher severity of fatigue.
Functional Assessment of Multiple Sclerosis (FAMS) Trial Outcome Index (TOI) at Year 11 | Year 11
  The Functional Assessment of Multiple Sclerosis (FAMS) instrument is a self-reporting, multi-dimensional, health-related QoL index for use in subjects diagnosed with MS. It comprised 58 items on 7 subscales (mobility, symptoms, emotional well-being, general contentment, thinking and fatigue, family/social wellbeing, and additional concerns). FAMS-TOI is the sum of the subscale scores mobility, symptoms, thinking/fatigue, and additional concerns. The items were rated on a 5-point scale (0 to 4). Score range of FAM-TOI is 0 to 148; the higher the score, the higher the quality of life. The evaluation period was the previous 7 days.
Functional Assessment of Multiple Sclerosis (FAMS) Total Score at Year 11 | Year 11
  The Functional Assessment of Multiple Sclerosis (FAMS) instrument is a self-reporting, multi-dimensional, health-related QoL index for use in subjects diagnosed with MS. It comprised 58 items on 7 subscales: mobility, symptoms, emotional well-being, general contentment, thinking and fatigue, family/social wellbeing, and additional concerns. The items were rated on a 5-point scale (0 to 4). Total score is sum of all sub-scale scores except 14 items for "Additional concerns", ranging 0 to 176; the higher the score, the higher the quality of life. The evaluation period was the previous 7 days.
PRO-based Efficacy Domain: European Quality of Life - 5 Dimensions (EQ-5D) Score at Year 11 | Year 11
  The EQ-5D measured five state-of-health dimensions: mobility, self-care, usual activities (work, leisure, etc.), pain/discomfort, and anxiety/depression. Every item had a score of 1 (no problems), 2 (some/moderate problems), or 3 (extreme problems). An individual's health status was defined in a combination of 5 digits. Subjects with missing answers to all questions were not considered for the respective visit.
European Quality of Life - 5 Dimensions (EQ-5D) Health-related quality of life (HRQoL) Score at Year 11 | Year 11
  Based on large population surveys, an algorithm was developed to combine the recordings of each of these five EQ-5D dimensions in 1 single HRQoL score, ranging from +1 (best imaginable HRQoL score) to -0.59 (worst imaginable HRQoL score). A relatively higher score represents better quality of life.
Number of Subjects who Started Second Line Therapy at Year 11 | Year 11
  Subjects were treated exclusively at the discretion of their treating physician and according to locally applicable standards and treatment guidelines. Subjects received second line therapy as a MS treatment such as alemtuzumab, cyclophosphamide, ciclosporin, fingolimod, methotrexate, mycophenolate mitoxantrone, natalizumab, etc.
Number of Subjects who Started First Disease-Modifying Treatment (DMT) other than IFNB at Year 11 | Year 11
  Subjects were treated exclusively at the discretion of their treating physician and according to locally applicable standards and treatment guidelines. All DMTs other than interferon beta, interferon beta-1a and interferon beta-1b were recorded as DMT other than IFNB.
Magnet-Resonance Imaging (MRI): Number of Newly Active Lesions | Year 11
  Contrast-enhanced MRI (with an extracellular gadolinium-based contrast agent) technique was used for the evaluation of brain lesions in MS. Newly active lesions defined as displaying either new enhancement on T1-weighted scans, or non-enhancing on T1-weighted scan but new on T2-weighted scans.
Magnet-Resonance Imaging (MRI): Number of Lesions on T1- and T2-Weighted Scans | Year 11
  Contrast-enhanced MRI (with an extracellular gadolinium-based contrast agent) technique was used for the evaluation of brain lesions in MS. Number of lesions on T1- and T2-Weighted scans were recorded.
Magnet-Resonance Imaging (MRI): Volume of Lesions on T1- and T2-Weighted Scans | Year 11
  Contrast-enhanced MRI (with an extracellular gadolinium-based contrast agent) technique was used for the evaluation of brain lesions in MS. Volume of lesions on T1- and T2-Weighted scans were recorded.
Magnet-Resonance Imaging (MRI): Normalized Brain Volume | Year 11
  Contrast-enhanced MRI (with an extracellular gadolinium-based contrast agent) technique was used for the evaluation of brain lesions in MS. Brain volume was analysed and reported.
Optical Coherence Tomography (OCT) Parameter - Retinal Nerve Fiber Layer (RNFL) | Year 11
  OCT is a noninvasive ocular imaging recognized in MS as a marker of axonal loss. Retinal nerve fiber layer (RNFL) thinning measured by OCT in subjects with MS occurs even in the absence of acute optic neuritis and is associated with worse scores for low-contrast letter acuity and other visual acuity tests. OCT measures peripapillary RNFL.
Optical Coherence Tomography (OCT) Parameter - Total Macular Volume (TMV) | Year 11
  OCT is a noninvasive ocular imaging recognized in MS as a marker of axonal loss. OCT is a potential method for capturing neuronal in addition to axonal degeneration in MS.
Optical Coherence Tomography (OCT) Parameter - Pupillo Macular Bundle (PMB) | Year 11
  OCT is a noninvasive ocular imaging recognized in MS as a marker of axonal loss. OCT is a potential method for capturing neuronal in addition to axonal degeneration in MS.
Optical Coherence Tomography (OCT) Parameter - Ganglion Cell Inner Plexiform Layer | Year 11
  OCT is a noninvasive ocular imaging recognized in MS as a marker of axonal loss. OCT is a potential method for capturing neuronal in addition to axonal degeneration in MS.
Ophthalmological examination - Optic Nerve Head | Year 11
  Standard clinical ophthalmic examination and test were applied for visual assessment and the differential diagnosis of OCT-related findings.
Ophthalmological examination - Slit lamp Biomicroscopy | Year 11
  Standard clinical ophthalmic examination and test were applied for visual assessment and the differential diagnosis of OCT-related findings. Ocular medical and surgical history, visual acuity (Early Treatment Diabetic Retinopathy Study Chart), low-contrast letter acuity (Sloan charts), and eye examination through slit-lamp biomicroscopy were assessed.
Ophthalmological examination - Visual Acuity | Year 11
  Standard clinical ophthalmic examination and test were applied for visual assessment and the differential diagnosis of OCT-related findings. Ocular medical and surgical history, visual acuity (Early Treatment Diabetic Retinopathy Study Chart), low-contrast letter acuity (Sloan charts), and eye examination through slit-lamp biomicroscopy were assessed.
Number of Subjects with Vitamin D Intake | Year 11
  Number of subjects with intake of Vitamin D were categorized as, 'since beginning of the BENEFIT study', and 'within the past 12 months'.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (75):
- Austria (2):
  - Graz, Styria
  - Innsbruck
- Belgium (4):
  - Bruxelles - Brussel
  - Ghent
  - Leuven
  - Liège
- Canada (4):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Brno
  - Hradec Králové
  - Ostrava-Poruba
  - Prague
- Glostrup Municipality, Denmark
- Finland (4):
  - Oulu
  - Seinäjoki
  - Tampere
  - Turku
- France (7):
  - Bordeaux
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Nice
  - Rennes
  - Toulouse
- Germany (16):
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Hennigsdorf, Brandenburg
  - Giessen, Hesse
  - Marburg, Hesse
  - Offenbach, Hesse
  - Göttingen, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Halle, Saxony-Anhalt
  - Erfurt, Thuringia
  - Münster
- Hungary (3):
  - Budapest
  - Debrecen
  - Szeged
- Israel (2):
  - Tel Litwinsky, Israel
  - Jerusalem
- Italy (6):
  - Orbassano, Torino
  - Gallarate
  - Milan
  - Padua
  - Pavia
  - Torino
- Sittard, Netherlands
- Bergen, Norway
- Poland (5):
  - Bydgoszcz
  - Krakow
  - Lodz
  - Lublin
  - Wroclaw
- Coimbra, Coimbra District, Portugal
- Ljubljana, Slovenia
- Spain (6):
  - Seville, Andalusia
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Madrid, Madrid
  - Málaga, Málaga
  - Valencia, Valencia
- Gothenburg, Sweden
- Switzerland (3):
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Sankt Gallen, Canton of St. Gallen
- United Kingdom (3):
  - Sheffield, South Yorkshire
  - Aberdeen
  - Dundee

REFERENCES:
- [Derived] Kappos L, Edan G, Freedman MS, Montalban X, Hartung HP, Hemmer B, Fox EJ, Barkhof F, Schippling S, Schulze A, Pleimes D, Pohl C, Sandbrink R, Suarez G, Wicklein EM; BENEFIT Study Group. The 11-year long-term follow-up study from the randomized BENEFIT CIS trial. Neurology. 2016 Sep 6;87(10):978-87. doi: 10.1212/WNL.0000000000003078. Epub 2016 Aug 10. PMID 27511182
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/